CLINICAL TRIAL: NCT03924505
Title: Preventing Opioid Overdose Mortality in the United States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Barrot Lambdin, Fellow, RTI International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INOD; R01DA046867 (NIH)
Record Dates: First submitted 2019-04-19; First posted 2019-04-23 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Opioid Overdose
Keywords: Implementation Science; Harm Reduction
MeSH Terms: conditions — Opiate Overdose; Harm Reduction | interventions — Organizations

STUDY DESIGN:
Masking Description: Study statistician was masked to which participants were in the intervention arm and which participants were in the control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organize and Mobilize for Implementation Effectiveness (Experimental): Our approach was based on the Implementation Sustainment Facilitation (ISF), which is grounded in the theory of implementation effectiveness, and added discrete strategies from the Addiction Technology Transfer Center (ATTC), which were considered necessary elements from the original ISF trial. In addition to receiving the OEND best practice recommendations, our multi-component approach used external facilitation as the overarching strategy, by which seven other strategies were leveraged to support SSP staff and leadership. In addition to external facilitation, the multi-faceted approach included: organize implementation team meetings, identify and prepare champions, develop and organize quality monitoring system, assess for readiness and identify barriers, distribute educational materials and resources, conduct educational meetings, and provide ongoing consultation.
  Interventions: Other: Organize and Mobilize for Implementation Effectiveness
- Dissemination of Best Practice Recommendations (Active Comparator): This arm will receive the best practice recommendations for implementing overdose education and naloxone distribution within syringe services programs.
  Interventions: Other: Dissemination

INTERVENTIONS:
Other: Organize and Mobilize for Implementation Effectiveness — Our trial is trying to understand how a multi-faceted, facilitation-based implementation strategy advances effective implementation of naloxone within syringe services programs
  Arms: Organize and Mobilize for Implementation Effectiveness
Other: Dissemination — Our comparison group receives dissemination of best practice recommendations for naloxone implementation.
  Arms: Dissemination of Best Practice Recommendations

SUMMARY:
This study aims to conduct a randomized controlled trial of 105 syringe services programs (SSPs) throughout the United States to understand the effectiveness of a multifaceted, facilitation-based strategy at advancing naloxone implementation effectiveness within SSPs. Together, these efforts can improve access to naloxone for people at high risk of overdose, thereby improving our nation's response to the opioid overdose epidemic.

DETAILED DESCRIPTION:
We conducted a randomized controlled trial of SSPs throughout the United States (US) and US Territories. Prior to the trial, 342 SSPs were known to be operating throughout the US and US Territories. Our team launched a national survey of syringe services programs (NSSSP) in February 2019 of all known SSPs operating throughout the United States and its Territories, receiving a response from 263 (77%) SSPs. Among the responding SSPs, 94% were implementing overdose education and naloxone distribution (OEND), and a total of 105 of SSPs implementing OEND were recruited into the trial. SSPs were randomized in a 1-to-1 fashion to either receive the OEND best practice recommendations (comparison SSPs) or the OEND best practice recommendations along with facilitation-based implementation strategies as detailed below (intervention SSPs).

We tested the effectiveness of a multifaceted, facilitation-based strategy at advancing OEND implementation effectiveness within SSPs. Implementation effectiveness is 'an organization-level construct that refers to the aggregated consistency, quality, and appropriateness of innovation use (OEND) within an organization (SSP).'

ELIGIBILITY:
To be eligible, an organization must have: 1) met the definition of an SSP - an organization whose primary function is to distribute drug use supplies to participants to reduce harms associated with drug use, 2) implemented OEND for a minimum of 6 months, and 3) completed the national survey of syringe services programs fielded February-July 2019. We excluded organizations such as fire departments or emergency departments of hospitals that offered supply distribution since it would be an ancillary function of these organizations and OEND programs that were not part of a syringe services program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barrot Lambdin, PhD, MPH, Principal Investigator — RTI International
Locations (1):
- RTI International, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lambdin BH, Bluthenthal RN, Garner BR, Wenger LD, Browne EN, Morris T, Ongais L, Megerian CE, Kral AH. Organize and mobilize for implementation effectiveness to improve overdose education and naloxone distribution from syringe services programs: a randomized controlled trial. Implement Sci. 2024 Feb 28;19(1):22. doi: 10.1186/s13012-024-01354-y. PMID 38419058

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: syringe services programs
Groups:
- Organize and Mobilize for Implementation Effectiveness: This arm will receive the naloxone intervention implementation manual and the External Facilitation (EF) intervention. The manual provides details for developing, implementing, and managing a naloxone intervention program within different types of organizations that serve people who use opioids, including SSPs. The EF intervention is a collaborative, organization-centered form of guiding to navigate barriers and leverage facilitators to advance an evidence-based intervention along the EPIS continuum. Guidance will be conducted by an External Facilitator.
  Implementation Manual with External Facilitation Intervention: Participating organizations will receive the implementation manual and the external facilitation (EF) intervention. The manual provides instructions for organizations wanting to implement a high quality naloxone program. The EF will assist syringe service programs to integrate naloxone delivery within their organization. As part of these efforts, we will use a measurement framework to understand naloxone delivery within SSPs along the four phases of the implementation process-exploration, preparation, implementation and sustainment (EPIS).
- Implementation Manual - Only: This arm will receive the naloxone intervention implementation manual. The manual provides details for developing, implementing, and managing a naloxone intervention program within different types of organizations that serve people who use opioids, including SSPs.
  Implementation Manual only: Participating organizations will receive the implementation manual.The manual provides instructions for organizations wanting to implement a high quality naloxone program.
Period: Overall Study
Arm/Group | Organize and Mobilize for Implementation Effectiveness | Implementation Manual - Only
Started | 53; 53 syringe services programs | 52; 52 syringe services programs
Completed | 51; 51 syringe services programs | 51; 51 syringe services programs
Not Completed | 2; 2 syringe services programs | 1; 1 syringe services programs

BASELINE CHARACTERISTICS:
Population: Our trial enrolled syringe services programs and randomized them to two arms. This was a study of organizations, not individuals.
Units Other Than Participants: Syringe Services Programs
Groups:
- Intervention Arm: This arm will receive the naloxone intervention implementation manual and the External Facilitation (EF) intervention. The manual provides details for developing, implementing, and managing a naloxone intervention program within different types of organizations that serve people who use opioids, including SSPs. The EF intervention is a collaborative, organization-centered form of guiding to navigate barriers and leverage facilitators to advance an evidence-based intervention along the EPIS continuum. Guidance will be conducted by an External Facilitator.
  Implementation Manual with External Facilitation Intervention: Participating organizations will receive the implementation manual and the external facilitation (EF) intervention. The manual provides instructions for organizations wanting to implement a high quality naloxone program. The EF will assist syringe service programs to integrate naloxone delivery within their organization. As part of these efforts, we will use a measurement framework to understand naloxone delivery within SSPs along the four phases of the implementation process-exploration, preparation, implementation and sustainment (EPIS).
- Control Arm: This arm will receive the naloxone intervention implementation manual. The manual provides details for developing, implementing, and managing a naloxone intervention program within different types of organizations that serve people who use opioids, including SSPs.
  Implementation Manual only: Participating organizations will receive the implementation manual.The manual provides instructions for organizations wanting to implement a high quality naloxone program.
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 53 | 52 | 105
Number analyzed (Syringe Services Programs) | 53 | 52 | 105
Age, Customized [Count of Participants; unit: Participants]
  Unknown | 53 | 52 | 105
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 35 | 31 | 66
  Male | 16 | 16 | 32
  Unknown/Not reported | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 45 | 38 | 83
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 8 | 9

OUTCOME MEASURES:

1. Primary Outcome: Naloxone Coverage (Consistency)
Description: Mean number of syringe services program participants receiving naloxone per total number of syringe services program participants
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: proportion of participants
Units Other Than Participants: syringe services programs
Groups:
- Organize and Mobilize for Implementation Effectiveness: Our approach was based on the Implementation Sustainment Facilitation (ISF) and added discrete strategies from the Addiction Technology Transfer Center (ATTC), which were considered necessary elements from the original ISF trial. In addition to receiving the OEND best practice recommendations, our multi-component approach used external facilitation as the overarching strategy, by which seven other strategies were leveraged to support SSP staff and leadership. These included: organize implementation team meetings, identify and prepare champions, develop and organize quality monitoring system, assess for readiness and identify barriers, distribute educational materials and resources, conduct educational meetings, and provide ongoing consultation.
  Regarding potential dose, SSP staff and organizational leadership were provided the opportunity to participate in 60-minute sessions once a month for up to 12 months. In addition to monthly sessions, facilitators were provided up to 2 hours to prepare for sessions and to identify and distribute resources to SSPs based on identified priorities. All sessions were offered virtually over audio-visual connections. Thus, the maximum possible dose for each SSP was 12 sessions or 36 hours.
- Dissemination of Best Practice Recommendations: Dissemination: Study staff disseminated best practice recommendations to all SSPs enrolled in the trial. To detail the OEND best practice recommendations, a Delphi study was carried out to develop a set of best practices for OEND implementation within SSPs. Experts for the Delphi study included people in paid and volunteer leadership and direct service positions in SSPs, OEND researchers, people who work in state or local health departments, and people who use drugs who deliver and access SSP/OEND services. All individuals had prior or current experience delivering OEND programming in community-based settings, and people with lived substance use experience were represented in each of the expert categories. Findings from this initiative were summarized into an organized best practices recommendations guide.
Arm/Group | Organize and Mobilize for Implementation Effectiveness | Dissemination of Best Practice Recommendations
Number analyzed (Participants) | 45 | 49
Number analyzed (syringe services programs) | 45 | 49
proportion of participants | 0.9 (1.4) | 0.4 (0.3)
Statistical Analysis 1: Comparison: Organize and Mobilize for Implementation Effectiveness vs Dissemination of Best Practice Recommendations; Test type: Superiority; p < 0.01, Negative Binomial Regression — A priori threshold for statistical significance set at p<0.05; We adjusted for baseline rate due to baseline differences; Incidence Rate Ratio = 2.15, 95% CI 2-sided [1.42 to 2.35] — The incidence rate ratio estimates the effect of facilitation for implementation effectiveness and dissemination of best practice recommendations, as compared to dissemination of best practice recommendations

2. Primary Outcome: Naloxone Doses Distributed (Consistency)
Description: The mean number of naloxone doses distributed per total number of SSP participants
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: naloxone doses
Units Other Than Participants: syringe services programs
Arm/Group | Organize and Mobilize for Implementation Effectiveness | Dissemination of Best Practice Recommendations
Number analyzed (Participants) | 46 | 50
Number analyzed (syringe services programs) | 46 | 50
naloxone doses | 2.5 (2.6) | 1.3 (1.2)
Statistical Analysis 1: Comparison: Organize and Mobilize for Implementation Effectiveness vs Dissemination of Best Practice Recommendations; Test type: Superiority; p = 0.01, Negative Binomial Regression — A priori threshold for statistical signicance is p<0.05; Incidence Rate Ratio = 1.97, 95% CI 2-sided [1.18 to 3.30] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Best Practice Adoption (Implementation Quality)
Description: The mean number of best practices adopted by the SSP
Time Frame: 12 months
Measure: Mean (Full Range); unit: number of best practices
Units Other Than Participants: syringe services programs
Arm/Group | Organize and Mobilize for Implementation Effectiveness | Implementation Manual - Only
Number analyzed (Participants) | 51 | 51
Number analyzed (syringe services programs) | 51 | 51
number of best practices | 13.1 [8 to 18] | 12.9 [8 to 17]
Statistical Analysis 1: Comparison: Organize and Mobilize for Implementation Effectiveness vs Implementation Manual - Only; Test type: Other — Testing for differences in means; p = 0.68, t-test, 2 sided; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.7 to 1.0], Standard Error of Mean 0.4

ADVERSE EVENTS:
Time Frame: 12 months of the intervention period
Description: Given that all of our interactions were with syringe service program staff/leadership, adverse events were only monitored at the syringe service program level and not at the syringe service program participant level.
Arm/Group | Organize and Mobilize for Implementation Effectiveness | Dissemination of Best Practice Recommendations
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 0/51 | 0/51

LIMITATIONS AND CAVEATS:
A noteworthy limitation with our trial is the reliance on self-report for the number of naloxone doses distributed, number of people receiving naloxone and best practice implementation. However, SSPs routinely report naloxone distribution metrics for funders. Generalizability of our study findings requires careful consideration. While we randomly selected SSPs to participate, it is possible that those that enrolled had different levels of resources than those that did not participate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT03924505/Prot_SAP_000.pdf